CLINICAL TRIAL: NCT04742855
Title: Effect of Probiotics on the Occurrence of Blepharitis in Adults and Children
Brief Title: Probiotics for Blepharitis in Adults and Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Other Study IDs: 01/2021
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Blepharitis
Keywords: microbiome/microbiota; probiotics
MeSH Terms: conditions — Blepharitis | interventions — Probiotics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: It will consist of 10 adults and 5 children. They will get the yogurt strains
  Interventions: Dietary Supplement: Probiotics
- Group B: It will consist of 10 adults and 5 children. They will get the Bifidobacterium strains.
  Interventions: Dietary Supplement: Probiotics
- Group C: It will consist of 10 adults and 5 children. They will get the placebo.

INTERVENTIONS:
Dietary Supplement: Probiotics — Study product is packaged as powders in a sachet. Participants and their parents will be instructed to dissolve the powder in water or milk, and to drink it in the morning and/or evening.
  Groups: Group A; Group B

SUMMARY:
The alteration of the intestinal microbiota through the use of specific probiotics can improve the clinical course of blepharitis by restoring intestinal and immune homeostasis. The purpose of this study is to define the possible positive impact of probiotics on patients with blepharitis.

DETAILED DESCRIPTION:
From recent studies, it has emerged that the gut microbiota is a possible responsible for the stimulation of the innate immune response and its role in the pathogenesis of autoimmune diseases has been deepened. Several clinical studies, in fact, support the existence of a connection between changes in the commensal intestinal microbiota ("dysbiosis") and autoimmune diseases. It has been seen that also ocular conditions like chalaziosis and uveitis are tied to dysbiosis. In addition, in a recent study probiotics were found to be safe and effective in the treatment of chalaziosis in children. Other eye conditions that may be affected by changes in the gut microbiome are dry eye syndrome and blepharitis. Under these conditions, a reduction in globet cells has often been noted. These cells produce the mucins present on the ocular surface, and therefore, their reduction involves the production of a thin and ineffective tear film. Therefore, the study will cover patients with blepharitis (both adults and children), treated with specific probiotics to be taken daily. Patients will then undergo a full ophthalmological examination each week for the first month, and then monthly until complete recovery for at least 6 months. In addition, at the time of enlistment and complete recovery, after venous sampling, the following biomarkers will be analyzed with cytometer and ELISA: TNFα and lymphocyte subpopulations. With this study, therefore, the aim is to define the possible positive impact of probiotics on patients with blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* blepharitis

Exclusion Criteria:

* eyelid infection
* suspicion of malignancy

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with blepharitis will be divided into three groups of 15 each (each group will be composed of 10 adults and 5 children)
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-01-18 (Estimated); Study Completion 2022-01-18 (Estimated)

PRIMARY OUTCOMES:
Blepharitis recurrence | six months
  assessment of the number of recurrences during the time frame of the study
Blepharitis resolution time | six months
  assessment of the number of days required for full resolution of the blepharitis

SECONDARY OUTCOMES:
systemic inflammatory profile | six months
  After venous sampling, the following biomarker will be analysed with a cytometer: TNFα (pg/mL) .
systemic inflammatory profile | six months
  After venous sampling, the following biomarker will be analysed with a cytometer: lymphocyte subpopulations (cells/mcL).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Molise, Campobasso, Italy

REFERENCES:
- [Result] Lu LJ, Liu J. Human Microbiota and Ophthalmic Disease. Yale J Biol Med. 2016 Sep 30;89(3):325-330. eCollection 2016 Sep. PMID 27698616
- [Result] Floyd JL, Grant MB. The Gut-Eye Axis: Lessons Learned from Murine Models. Ophthalmol Ther. 2020 Sep;9(3):499-513. doi: 10.1007/s40123-020-00278-2. Epub 2020 Jul 2. PMID 32617914
- [Result] Moon J, Yoon CH, Choi SH, Kim MK. Can Gut Microbiota Affect Dry Eye Syndrome? Int J Mol Sci. 2020 Nov 10;21(22):8443. doi: 10.3390/ijms21228443. PMID 33182758
- [Result] Filippelli M, dell'Omo R, Amoruso A, Paiano I, Pane M, Napolitano P, Bartollino S, Costagliola C. Intestinal microbiome: a new target for chalaziosis treatment in children? Eur J Pediatr. 2021 Apr;180(4):1293-1298. doi: 10.1007/s00431-020-03880-5. Epub 2020 Nov 23. PMID 33226501
- [Result] Ochoa-Reparaz J, Kasper LH. The influence of gut-derived CD39 regulatory T cells in CNS demyelinating disease. Transl Res. 2017 Jan;179:126-138. doi: 10.1016/j.trsl.2016.07.016. Epub 2016 Jul 28. PMID 27519147
- [Result] Cavuoto KM, Banerjee S, Galor A. Relationship between the microbiome and ocular health. Ocul Surf. 2019 Jul;17(3):384-392. doi: 10.1016/j.jtos.2019.05.006. Epub 2019 May 21. PMID 31125783
- [Result] Moon J, Choi SH, Yoon CH, Kim MK. Gut dysbiosis is prevailing in Sjogren's syndrome and is related to dry eye severity. PLoS One. 2020 Feb 14;15(2):e0229029. doi: 10.1371/journal.pone.0229029. eCollection 2020. PMID 32059038